CLINICAL TRIAL: NCT06459063
Title: A Placebo-controlled Study of Intra-articular Allocetra in Osteoarthritis of the 1st Carpo-metacarpal Joint
Brief Title: Intra-articular Allocetra in Osteoarthritis of the 1st Carpo-metacarpal Joint
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Amir Oron, MD, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0006-24-KMC
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis Thumb
Keywords: Allocetra; Cell therapy; Carpo-metacarpal; Osteoarthritis; Thumb; Macrophage
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety run-in phase - Allocetra increasing dose (Other): A dose escalation phase to characterize the safety of Allocetra injection to the 1st CMC joint in the target thumb in different doses and select the dose for the randomized phase.
  Interventions: Drug: Allocetra - Safety run-in phase
- Randomization phase - Allocetra (Active Comparator): Injection of Allocetra to the 1st CMC joint in the target thumb.
  Interventions: Drug: Allocetra - Randomization phase
- Randomization phase - Placebo (Placebo Comparator): Injection of placebo to the 1st CMC joint in the target thumb.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Allocetra - Safety run-in phase — Intra-articular injection of Allocetra performed once on Day 1 of the study at different doses.
  Arms: Safety run-in phase - Allocetra increasing dose
Other: Placebo — Intra-articular injection of placebo solution containing all excipients except for the Allocetra cells.
  Arms: Randomization phase - Placebo
Drug: Allocetra - Randomization phase — Intra-articular injection of selected dose of Allocetra based on the safety run-in, performed on Day 1 of the study.
  Arms: Randomization phase - Allocetra

SUMMARY:
This study is a single center trial to assess the safety and efficacy of intra-articular administration of Allocetra to patients with 1st CMC thumb joint osteoarthritis (OA).

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the first carpometacarpal (CMC) joint, or basal joint of the thumb, is a common, painful, and debilitating disease. For patients whose symptoms persist despite conservative therapies and rehabilitation strategies, surgery remains the last-resort treatment.

Allocetra is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

This study is a single center safety and efficacy assessment trial to assess intra-articular administration of Allocetra in patients suffering from thumb osteoarthritis in the 1st CMC joint (basal thumb joint) who have not responded sufficiently to conventional therapies.

The study is comprised of a safety run-in stage to characterize safety of Allocetra injections at different doses, followed by a placebo-controlled double-blind randomized stage to evaluate the safety and efficacy of Allocetra injection to the basal thumb joint.

Patients will be followed for up to a year following treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this clinical study must fulfill all of the following:

1. Age 40 years or older.
2. Patients with OA of the first CMC joint of the target thumb (basal thumb joint) who have failed conventional therapies, with pain assessed when not taking analgesic medications.
3. Score of 6 or higher on the Functional Index for Hand Osteoarthritis (FIHOA).
4. X-ray confirming OA of the first CMC joint of the target thumb with a Grade of 2 or 3 according to Eaton classification.
5. Blood tests from up to three months before treatment within protocol-defined limits.

Exclusion Criteria:

Subjects not eligible for this study include those that have any of the following:

1. Any significant injury, fracture, surgery, active local infection, deformity, severe Carpal Tunnel Syndrome (CTS), DeQuervain's tenosynovitis, trigger finger, or a ganglion cyst of the target hand.
2. History of chondrocalcinosis in the target joint, concomitant rheumatic disease.
3. Previous intra-articular injection of steroid, hyaluronate, or other agent, into the target joint within 3 months prior to screening visit.
4. Other limb pain of unknown etiology, or clinically significant widespread pain syndrome, e.g., fibromyalgia.
5. Pain in the limb clinically assessed to arise from an origin which is not the affected thumb joint (wrist pain, shoulder pain, etc.).
6. Secondary OA such as gout, hemochromatosis, rheumatoid/psoriatic arthritis.
7. Bleeding disorders, cognitive disorder, neurologic disease or other major medical condition which may interfere with study participation, treatment, assessments, or results.
8. For women of childbearing potential, a positive pregnancy test.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Injection-related reactions | Day 0 (Treatment visit).
  Injection-related reactions occurring during study treatment injection, including injection interruption/discontinuation.
Treatment emergent adverse events | Day 0 to 6 months.
  Treatment emergent adverse events following study treatment injection. Safety assessments beyond 4 weeks following injection will focus on events that are at least possibly related to study treatment.

SECONDARY OUTCOMES:
Thumb base pain - NRS | Screening day to 12 months.
  Thumb base pain numerical rating scale (NRS; 0-10).
Hand function - FIHOA | Day 0 to 12 months.
  Hand function, assessed by Functional Index for Hand Osteoarthritis (FIHOA; 0-30).
Key pinch and grip strength | Day 0 to 12 months.
  Key pinch and grip strength - measured with dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

REFERENCES:
- [Background] Armstrong AL, Hunter JB, Davis TR. The prevalence of degenerative arthritis of the base of the thumb in post-menopausal women. J Hand Surg Br. 1994 Jun;19(3):340-1. doi: 10.1016/0266-7681(94)90085-x. PMID 8077824